CLINICAL TRIAL: NCT07056049
Title: Efficacy of High-dosage, High-intensity Rehabilitation Program on the Motor Recovery After Stroke in Subacute Patients
Brief Title: The Efficacy of Additional Motor Training Dosage During the Early Stages Post Stroke on the Upper Extremity Recovery
Acronym: EFODIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adi Negev-Nahalat Eran (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGV-24-0006
Record Dates: First submitted 2025-06-10; First posted 2025-07-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Hemiplegia and Hemiparesis
Keywords: Stroke Rehabilitation; Motor Impairment; Post-stroke High Dosage Rehab; Technological Rehab Post Stroke; Stroke Kinematics
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis

STUDY DESIGN:
Intervention Model Description: The intervention group will be compared to a matched historical cohort, that will be added to in parallel during recruitment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This group will be provided with additional rehab time during the sub actue phase. (Experimental): Participants will receive additional technology-based upper extremity training for 120 min/day, 5d/w, 4 weeks.
  The program will be tailored to their impairment level, and will be added to the usual treatment given during hospitalization.
  Interventions: Behavioral: High dosage, high intensity motor rehabilitation
- Matched group from an ongoing project with identical criteria. (No Intervention): This group is comprised of patients with similar characteristics and the intervention group will be compared to this group.

INTERVENTIONS:
Behavioral: High dosage, high intensity motor rehabilitation — Participants will receive additional technology-based upper extremity training for 120 min/day, 5d/w, 4 weeks.
  Arms: This group will be provided with additional rehab time during the sub actue phase.

SUMMARY:
Intervention abstract

Background: Stroke is the leading cause of long-term disability, and the second leading cause of death in the western world. Most stroke survivors will suffer from motor and cognitive disturbances for the rest of their life, which negatively affects their normal daily life.

Despite the decline in stroke-related mortality over the past decades, the outcome of rehabilitation programs does not improve, and is predictable regardless of the program used. Still, several human and animal studies show that high capacity of training in the early stages post stroke improve motor recovery. This notion is far from being well established.

Aim: Studying the effect of high-dosage, high-intensity training program in the subacute period on upper extremity motor recovery.

Population: Stroke survivors. Study duration: 6 months. Study protocol: Participants will receive additional technology-based upper extremity training for 120 min/day, 5d/w, 4 weeks. They will be monitored pre and post training, and 6 months post-stroke. Outcome measures will include clinical, kinematic and adherence measures (see complete list in the protocol).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ischemic or hemorrhagic stroke (hemispheric or brainstem) confirmed by CT or MRI
* First-ever stroke or previous stroke with no upper extremity weakness
* 1 week ≤ Time after stroke onset ≤ 6 weeks
* Active shoulder flexion of at least 20◦ and partial wrist and/or finger active movement
* Ability to provide inform consent

Exclusion Criteria:

* A painful shoulder limiting an active forward reach
* Severe spasticity or non-neural loss of range of motion
* Cognitive or communication impairments as determined by the clinical team Unstable medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer upper extremity assessment (FM-UE) | Enrollment, 1 month, 3 months, 6 months after enrollment
  The Upper Extremity Fugl-Meyer Assessment (UE-FMA) is a standardized clinical tool designed to evaluate motor impairment in the upper limb following a stroke. It is part of the broader Fugl-Meyer Assessment, one of the most widely used and validated scales in stroke rehabilitation research. The UE-FMA specifically assesses movement, coordination, and reflexes in the shoulder, elbow, forearm, wrist, and hand, with a maximum score of 66 points. The scale is divided into subcomponents, including upper limb movement (36 points), wrist (10 points), hand (14 points), and coordination/speed (6 points). Each item is scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully), offering a total score that reflects the level of motor impairment-higher scores indicate better motor function. The UE-FMA is valued for its reliability, sensitivity to impairment (rather than function), and its ability to track motor recovery over time.
Action research arm test (ARAT) | Enrollment, 1 month, 3 months, 6 months after enrollment
  The Action Research Arm Test (ARAT) is a standardized clinical tool used to assess upper limb function following stroke or neurological injury, with a focus on evaluating the ability to perform purposeful, goal-directed tasks. It consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement, each designed to measure different aspects of upper limb activity. Tasks include actions such as picking up small blocks, pouring water, or moving objects across a table. Each item is scored on a 4-point ordinal scale ranging from 0 (no movement) to 3 (normal performance), yielding a maximum total score of 57. The ARAT captures the functional use of the hand and arm in a way that reflects real-world tasks, making it especially relevant for tracking meaningful improvements during rehabilitation. It is known for its high inter-rater and intra-rater reliability and is sensitive to changes in functional performance across a wide spectrum of impairment levels.
Stroke Impact Scale (SIS) hand domain, version 2.0 | Enrollment, 1 month, 3 months, 6 months after enrollment
  The Stroke Impact Scale (SIS) hand domain, version 2.0, is a patient-reported outcome measure that assesses the perceived difficulty of using the affected hand in everyday tasks following a stroke. This domain includes five items that ask individuals to rate the difficulty of performing common activities such as carrying heavy objects, turning a doorknob, or picking up a coin. Each item is scored on a 5-point Likert scale ranging from 1 (could not do it at all) to 5 (not difficult at all), reflecting the patient's experience over the past week. Scores are converted to a 0-100 scale, with higher scores indicating better perceived hand function. The SIS hand domain captures the individual's perspective on the functional impact of stroke on daily activities, providing valuable insight into real-world hand use. It is frequently used in stroke rehabilitation studies to complement performance-based assessments and to evaluate patient-centered outcomes.
Kinematics | Enrollment, 1 month, 3 months, 6 months
  Using reaching tasks that will be recorded using multiple high resolution video-cameras and analyzed using AI algorithm (OpenPose). Outcome measures that will be examined include: trajectory smoothness, reaching extent, shoulder-elbow synergy, movement time and deviation from trajectories of age matched healthy controls.

SECONDARY OUTCOMES:
Upper extremity activity | Enrollment and 3 months.
  Daily natural activity will be monitored for using IMUs (Movella DOT) worn on upper extremity and trunk for periods of up-to 6 hours.
Time on task | The measure will be recorded every single practice session, twice a day, 5 days a week. Total Time on Task will be calculated at the end of the intervention period, approximately 4 weeks.
  Actual time spent training during a practice session.
Attendance | The measure will be recorded every single practice session, twice a day, 5 days a week. Total attendance will be calculated at the end of the intervention period, approximately after 4 weeks.
  The rate in which a participant actively participated in the training sessions.
Visual Analogue Scale for pain | The measure will be recorded before and after every single practice session, twice a day, 5 days a week. The mean pain level delta will be calculated at the end of the intervention period, approximately 4 weeks.
  The VAS is a self-report measure consisting of a 10 centimeter line with a statement at each end representing one extreme of pain intensity (No pain and pain as bad as it could possibly be). The participant gives their indication with a pen mark on the line corresponding to their present pain level. The higher the score, the worse the pain.
Rating of perceived exertion (RPE) | The measure will be recorded every single practice session, twice a day, 5 days a week.
  The revised category-ratio scale (0 to 10 scale) will be used to monitor and guide exercise intensity. Participants subjectively rate their level of exertion during exercise (American College of Sports Medicine, 2010). A higher score means higher exertion experienced by the participant during the session.
  It is not necessarily good or bad, it is just an indication of the effort.
The Intrinsic Motivation Inventory (IMI) | At the end of the intervention period for each participant (i.e. 4 weeks).
  The IMI is a validated self-report tool used to assess intrinsic motivation toward a specific activity. It includes multiple subscales, with Interest/Enjoyment considered the primary indicator of intrinsic motivation. Items are rated on a 7-point Likert scale (1 = not at all true, 7 = very true), and subscale scores are averaged to produce interpretable values. Higher scores reflect greater intrinsic motivation, perceived competence, or effort, depending on the subscale.

OTHER OUTCOMES:
Berg Balance Scale (BBS) | Only at enrollment.
  Consists of 14 items for assessing static and dynamic balance and risk of falls for different populations. The test includes different tasks in various challenging positions and scored up to 56 points. A higher score indicated better balance and lower risk of falls.
Fatigue Severity Scale (FSS) | At the end of the intervention period (i.e. 4 weeks)
  The 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. A higher scale indicated higher fatigue level.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Shmuelof, Prof., Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Adi Negev-Nahalat Eran, Ofakim, Israel

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data to be shared will include de-identified information collected during the trial, such as demographic and baseline characteristics, intervention allocations, and all outcome measures used in both the primary and secondary analyses. In addition, supporting documentation will be provided to facilitate proper use of the data, including the study protocol, statistical analysis plan, informed consent form template, and a comprehensive data dictionary.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The de-identified individual participant data and supporting documentation will be made available beginning six months after publication of the primary results and will remain accessible for a minimum of five years thereafter.
Access Criteria: Qualified researchers with a scientifically sound proposal will be able to request access to the de-identified individual participant data and supporting documents, including the study protocol, statistical analysis plan, informed consent form template, and data dictionary. Access will be granted through a secure data repository following submission and approval of a data access request. Researchers will be required to sign a data use agreement outlining conditions for responsible data use, including maintaining confidentiality and using the data only for the approved purpose. Access will be provided through controlled mechanisms, such as registered user accounts or institutional credentials, depending on the repository's access procedures.

REFERENCES:
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Background] Buch ER, Rizk S, Nicolo P, Cohen LG, Schnider A, Guggisberg AG. Predicting motor improvement after stroke with clinical assessment and diffusion tensor imaging. Neurology. 2016 May 17;86(20):1924-5. doi: 10.1212/WNL.0000000000002675. Epub 2016 Apr 29. No abstract available. PMID 27164664
- [Background] Biernaskie J, Chernenko G, Corbett D. Efficacy of rehabilitative experience declines with time after focal ischemic brain injury. J Neurosci. 2004 Feb 4;24(5):1245-54. doi: 10.1523/JNEUROSCI.3834-03.2004. PMID 14762143